CLINICAL TRIAL: NCT03379233
Title: A 24-week Randomized, Controlled, Multicenter, Open-label Study to Evaluate the Effect of Reminder Notifications and Motivational/Adaptive Messaging on Treatment Adherence of COPD Subjects Receiving Ultibro® Breezhaler® Treatment Using the Concept2 Inhaler for Dose Administration and Tracking
Brief Title: A Randomized Study to Evaluate the Effect of Reminder Notifications and Motivational/Adaptive Messaging on Treatment Adherence
Acronym: ADVICE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: devices malfunctioned
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIDD001D2402
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Adherence; Dose Tracking; Concept2; Digital Adherence System; Ultibro Breezhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Concept2 inhaler
  Interventions: Combination Product: Concept2 inhaler
- Telehealth (Experimental): Concept2 inhaler with patient application
  Interventions: Combination Product: Concept2 inhaler with patient application

INTERVENTIONS:
Combination Product: Concept2 inhaler — Fixed combination of Indacaterol maleate (QAB149) and glycopyrronium bromide (NVA237), 110/50 μg, capsule added to Concept2 inhaler
  Arms: Usual Care
Combination Product: Concept2 inhaler with patient application — Fixed combination of Indacaterol maleate (QAB149) and glycopyrronium bromide (NVA237), 110/50 μg, capsule added to Concept2 inhaler with application used for monitoring
  Arms: Telehealth

SUMMARY:
This study was evaluating the effect of reminder notifications and motivational/adaptive messages on treatment adherence behavior in subjects with COPD. The effect will be measured over 24 weeks on the subject's on time treatment adherence and total treatment adherence. The delivery of the medication and tracking of inhaler use is done by the Concept2 inhaler. The reminder notification, feedback on inhaler use and motivational messages are provided by the patient application, who is receiving the inhaler use information from the Concept2 inhaler.

DETAILED DESCRIPTION:
This study was evaluating whether subjects with COPD on Ultibro® Breezhaler® clinical trial formulation once daily dosing regimen using the Concept2 inhaler in conjunction with a patient application collecting data and sending reminder notifications and motivational/adaptive messages aimed at encouraging treatment adherence, have improved treatment adherence compared to subjects using the Concept2 inhaler alone (usual care). The delivery of the medication and tracking of inhaler use is done by the Concept2 inhaler. The reminder notifications, feedback on inhaler use and motivational messages for the subject are sent by the patient application based on the received subjects inhaler use information from the Concept2 inhaler.

The effect will be measured over 24 weeks on the subject's on time treatment adherence (days when the subjects inhaled within +/- 2 hours of the subjects preferred inhalation time) and total treatment adherence (days when patient inhaled at least one dose).

The study population consisted male and female adult patients, 18 years or older with a clinical diagnosis of COPD, a smoking history of 10 pack years, receiving Ultibro Breezhaler treatment for at least 3 months prior to screening and documented poor treatment adherence.

After 6 weeks of screening patients will be randomized to either the Usual Care group in which they will continue to receive Ultibro Breezhaler treatment via the Concept2, or the Telehealth group in which they will additionally receive a tablet device pre-installed with a patient app.

In addition to on time treatment adherence and total treatment adherence, illness and treatment beliefs will be collected via a questionnaire and patient's health status from the EQ5D-5L and SGRQ-C Questionnaire. Key safety assessments are COPD exacerbation and AE/SAE, device deficiencies and device events, drug administration errors, physical exam, vital signs and urine or serum pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Have a total adherence of more than 10% but less than or equal to 70% during Screening period
* Current or ex-smokers who have a smoking history of at least 10 pack years.
* A diagnosed COPD
* Taking Ultibro® Breezhaler® for at least 3 month prior to Visit 1
* Have been in the Screening period ≥ 35 days.

Exclusion Criteria:

* Pregnant or lactating women
* Women of child-bearing potential
* Subjects having a history of reactions/hypersensitivity to inhaled drugs or drugs of a similar class
* Subjects having a history of reactions/hypersensitivity to lactose or any of the other ingredients of trial medication.
* Subjects with relevant concomitant diseases
* Subjects who have had a COPD exacerbation 6 weeks prior to Visit 1 or between V1 and randomization
* Subjects who have had a respiratory tract infection within 3 weeks prior to Visit 1 or between V1 and randomization
* Use of investigational drugs or other investigational devices at the time of enrollment
* Subjects with a preferred inhalation time between 10.00 pm and 2.00 am.
* Subjects taken off Ultibro® Breezhaler® treatment/inhaler use by the investigator during the Screening period for more than 7 days.
* Subjects not returning all Concept2 inhalers received during the Screening period
* Subjects who have demonstrated inability or unwillingness to use the digital system or to fill in questionnaires.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
- Netherlands (4):
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Helmond
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Zutphen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Netherlands and Germany between 11 July 2018 (first participant first visit) and 22 January 2019 (last participant last visit).
Pre-assignment Details: A total of 7 subjects were randomized in the study.
Groups:
- Telehealth Group: Participants inhaled Ultibro Breezhaler 110/50 micrograms (mcg) clinical formulation once daily via Concept2 inhaler with an electronic connectivity to a patient application pre-installed on a tablet device for 24 weeks.
- Usual Care Group: Participants inhaled Ultibro Breezhaler 110/50 mcg capsule once daily via Concept2 inhaler for 24 weeks.
Period: Overall Study
Arm/Group | Telehealth Group | Usual Care Group
Started | 1 | 6
Completed | 0 | 0
Not Completed | 1 | 6
Not completed — Technical issues with Concept 2 inhalers | 1 | 6

BASELINE CHARACTERISTICS:
Population: Randomized set consisted of all participants who were randomized to one of the interventions (Telehealth group or Usual Care group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Telehealth Group | Usual Care Group | Total
Number analyzed (Participants) | 1 | 6 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 6 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 6 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 1 | 2 | 3
  Germany | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Participant's On-time Adherence Over 24 Weeks of Intervention Compared to Baseline
Description: On-time treatment adherence was defined as percentage of days on which the participant inhaled at least one dose on-time. Dose inhaled on-time was a dose inhaled within (+ or -) 2 hours of the agreed predefined preferred daily inhalation time (PIT). PIT was defined by the participant at study start.
Time Frame: Baseline 6 weeks, intervention 24 weeks
Population: Due to technical issues, the actual time and day of inhaler use from the point of resetting could not be evaluated. Therefore data for this outcome measure were not collected and reported.
Arm/Group | Telehealth Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Participant's Total Adherence Over 24 Weeks of Intervention Compared to Baseline
Description: Total adherence was defined as percentage of days on which the participant inhaled at least one dose and represented the sum of on-time adherence and off-time adherence. Off-time adherence was defined as percentage of days on which the participant did not inhale the daily dose within the (+ or -) 2 hours of the predefined PIT, but outside. The number of doses not inhaled on-time was recorded by the Concept2 inhaler.
Time Frame: Baseline 6 weeks, intervention 24 weeks
Population: as for outcome 1
Arm/Group | Telehealth Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Participant's 6 Weeks Baseline On-time Adherence to the Participant's On-time Adherence Over the Last Four Weeks of Intervention
Description: as for outcome 1
Time Frame: Baseline, Week 21 - 24
Population: Due to the early discontinuation of the study, only very few participants were randomized (7) and no participant completed the last 4 weeks of intervention, required for the evaluation of the secondary efficacy outcome measure. Therefore data for this outcome measure was not collected and reported.
Arm/Group | Telehealth Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Participant's 6 Weeks Baseline Total Adherence to the Participant's Total Adherence Over the Last Four Weeks of Intervention
Description: as for outcome 2
Time Frame: Baseline, Week 21 - 24
Population: as for outcome 3
Arm/Group | Telehealth Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were reported from start of treatment up to follow up (34 weeks)
Description: Enrolled set consisted of participants who signed informed consent and had some assessment done in the screening period.
Arm/Group | Telehealth Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/6
Other Adverse Events (participants affected / at risk) | 0/1 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telehealth Group (N=1) | Usual Care Group (N=6)
Respiratory tract infection (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to technical issues with the investigational Concept2 inhalers. Due to limited and inaccurate data, efficacy endpoints with respect to change in on-time and total treatment adherence were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT03379233/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT03379233/SAP_001.pdf